CLINICAL TRIAL: NCT01110278
Title: Examining the Brain's Control Systems in Normal and Overactive Bladder Using DTI and Functional MRI
Brief Title: Examining Bladder Control Using Magnetic Resonance Imaging (MRI) and Diffusion Tensor Imaging (DTI)
Status: Completed | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Rahel Nardos, MD, Oregon Health and Science University
Other Study IDs: OHSU eIRB 6005
Record Dates: First submitted 2010-04-16; First posted 2010-04-26 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Urinary Incontinence, Urge
Keywords: Urge Urinary Incontinence; Magnetic Resonance Imaging; Diffusion Tensor Imaging; Brain Connectivity; Bladder Control; fMRI
MeSH Terms: conditions — Urinary Incontinence, Urge

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Urge Incontinent Women: Women with documented urge/urgency incontinence with established care at the Oregon Health and Science University.
- Control Women: Women with no urge/urgency incontinence with established care at the Oregon Health and Science University.

SUMMARY:
Urgency incontinence (where the bladder muscles contract suddenly, causing an immediate urge to urinate that is difficult to prevent) is commonly experienced in patients with overactive bladder. New findings have discovered that urgency incontinence may be connected to the interactions of certain regions of the brain and the bladder. Although this is a common problem, researchers still do not know how these interactions impact the process of urgency incontinence. The purpose of this study is to better understand how the brain functions, by using Magnetic Resonance Imaging (MRI) machine and Diffusion Tensor Imaging (DTI) to create images of the brain during different bladder states.

DETAILED DESCRIPTION:
One devastating manifestation of overactive bladder is urgency incontinence. Although urgency incontinence is a common problem with profound clinical, social and psychological consequences, little is understood about its underlying cause. The involuntary detrusor overactivity (DO) often associated with the disease points to a possible abnormality in voluntary control of the spinobulbospinal voiding reflex by a higher order neuronal network. Recent functional MRI (fMRI) and PET studies have identified increased brain activity during bladder filling and voiding in normal subjects from higher order cognitive control centers. In addition, there are now data to suggest that interactions between these brain areas, which include the pontine micturition center (PMC), periaqueductal gray (PAG), thalamus, insula, dorsal anterior cingulate and prefrontal cortex, may be abnormal in patients with urgency incontinence. Despite these encouraging findings, we do not yet know how these regions are interacting with each other, or to other, unknown but important, regions in the brain. Nor do we know how this interaction might play a role in this disease process. Expanding our knowledge of how these regions are integrated to achieve continence and, importantly, what aspects of this complex circuitry are atypical in patients with urge incontinence is key to our future therapeutic endeavors. With this in mind, the goal of this study is to better characterize the functional integration (i.e. functional connectivity) of the brain's control networks in relation to typical and atypical bladder function. We aim to identify distinct differences in the brain's functional and anatomic topography in women with and without urgency incontinence. Our approach not only has the potential to advance our understanding of the higher level pathophysiology of this disease process, but could also lead to novel more centrally acting therapeutic approaches for treatment of urgency incontinence.

ELIGIBILITY:
CASE GROUP: This group will include 15 patients presenting to the urogynecology clinic at OHSU with current bladder overactivity symptoms including urgency and urgency incontinence with documented detrusor overactivity on multichannel urodynamic assessment.

Inclusion criteria:

* Female urogynecology patients between age 40 and 85.
* Without a history of incontinence surgery
* Have current overactive bladder symptoms including urgency and urgency incontinence daily for the previous three months (must answer "about once a day to Question A1:how often do you leak urine, on initial screening questionnaire, and "3 or more months to question A2: How long have you experienced accidental leakage, and "yes" to question A3:Do you usually experience urinary leakage associated with feeling of urgency).
* Documented detrusor overactivity by urodynamic study within 3 months of the study is required.
* Patients who have a history of past anticholinergic therapy will be included as long as they have been off medication for 2 weeks prior to imaging.

Exclusion criteria:

* Medical contraindications for MRI scanning.
* Past or present overt neurological disease such as history of stroke, epilepsy, MS, spinal cord injury.
* History of pelvic irradiation or bladder cancer.
* Current urinary tract infection.
* Current pelvic pain disorder.

CONTROL GROUP: This group will include 25 gynecology patients without a history of any urinary incontinence symptoms.

Inclusion Criteria:

* Female gynecology patients between age 40 and 85.
* Without a history of urinary incontinence (must answer "never" to question A1: how often do you leak urine, on initial screening questionnaire).
* Without a history of incontinence surgery.
* Without a history of overactive bladder.
* Without pelvic pain.
* Without irritative bladder symptoms (must say "no" to question A4: do you experience frequent urination on initial screening questionnaire).

Exclusion criteria:

* Medical contraindications for MRI scanning.
* Past or present overt neurological disease such as history of stroke, epilepsy, MS, spinal cord injury.
* History of pelvic irradiation or bladder cancer.
* Current urinary tract infection.
* Current pelvic pain disorder.

Ages: 40 Years to 85 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women seeking care at Oregon Health and Science University in Portland, Oregon.
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2010-05; Primary Completion 2012-06-22 (Actual); Study Completion 2012-06-22 (Actual)

PRIMARY OUTCOMES:
Determine differences in fluctuations in brain activity between different regions of the brain associated with control functions. | Once during up to 3 months
  We will look at the overall group differences to see if there are differences between the case group participants and control group participants in control brain regions related to normal bladder function.

SECONDARY OUTCOMES:
Scores on the Pelvic Floor Distress Inventory | Once during up to 3 months
  This Questionnaire is a condition-specific quality of life questionnaire to assess pelvic floor disorders including urinary incontinence, pelvic organ prolapse and fecal incontinence.
3 Day Bladder Diary to Assess Participant Symptom Severity | Once during up to 3 months
  Subjects will be given three questionnaires and will also be asked to keep a diary that tracks their bladder and urinary habits for 3 days.
Determine any difference in brain response to bladder filling in subjects with and without overactive bladder. | Once during up to 3 months
Determine functional brain connectivity with bladder. | Once during up to 3 months
  In order to asses functional connectivity (measurement of the strength of integration between brain regions), direct statistical comparison of connectivity maps derived from urge incontinence versus control groups will be done.
Scores on the Pelvic Floor Impact Questionnaire | Once during up to 3 months
  This is another validated brief quality of life questionnaire to assess how various pelvic floor disorders affect specific daily activities.
Scores on the International Consultation on Incontinence Questionnaire | Once during up to 3 months.
  This questionnaire allows assessment of the prevalence, frequency and perceived cause of urinary incontinence as well as its impact on life.

CONTACTS AND LOCATIONS:
Overall Officials: Rahel Nardos, M.D., Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States